CLINICAL TRIAL: NCT04397640
Title: Study of Myocardial Microcirculatory Alterations in Patients With Sepsis and Septic Shock Using Myocardial Contrast Echocardiography (MCE)
Brief Title: Myocardial Contrast Echocardiography in Septic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Duc Nam Nguyen, Clinical Professor, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN 3202042835
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Sepsis; Microcirculation
Keywords: Sepsis; Septic cardiomyopathy; Contrast echocardiography; Sulphur hexafluoride microbubbles contrast Sonovue
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Cohort study in a single center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonovue (Other): ICU patients with sepsis and septic shock who are eligible for myocardial contrast echocardiography with sulphur hexafluoride microbubbles contrast Sonovue (Bracco, Milan, Italy) injection.
  Interventions: Diagnostic Test: Sonovue

INTERVENTIONS:
Diagnostic Test: Sonovue — Contrast myocardial echocardiography with sulphur hexafluoride microbubbles Sonovue (Bracco, Milan, Italy) injection and using the time-intensity curves profile to evaluate the myocardial microcirculation.

SUMMARY:
Myocardial microcirculatory alterations may be involved in the pathogenesis of acute cardiac dysfunction or septic cardiomyopathy in septic patients. The investigators study the cardiac function (systolic and diastolic) with two-dimensional echocardiography (TTE), and the myocardial microcirculation with contrast echocardiography (MCE) and sulphur hexafluoride microbubbles Sonovue injection in ICU septic patients.

DETAILED DESCRIPTION:
Using the IE33 device (Philips Medical Systems, the Netherlands), two-dimensional and myocardial contrast echocardiography (TTE and MCE) are performed following the recommendations of the American Heart Association and the European Society of Cardiology (2006), and the European Association of Cardiovascular Imaging (2017). TTE and MCE are performed at the same time in the first 24 hours after ICU admission, at 48-72 hours, at 5-10 days after withdrawal of vasopressors and inotropes.

First, TTE evaluates from the apical and parasternal views:

* The Wall motion score index (WMSI) of 16 myocardial segments of the left ventricle (LV).
* The diastolic function using pulsed-wave doppler and pulsed tissue doppler at the mitral valve.
* Quantify valvular insufficiency
* Estimation of cardiac output (L/ minute).
* Evaluation of the right ventricle (RV) dimension and its the longitudinal contractility by the Tricuspid annular plane systolic excursion (TAPSE) with pulsed tissue doppler.
* Left atrial volume (ml).
* Systolic pulmonary pressure and pulmonary resistance with both continuous and pulsed-wave doppler at the tricuspid valve and the pulmonary outflow tract, respectively.

Second, MCE is performed if:

* Systolic blood pressure < 200 mmHg or > 90 mmHg,
* Heart rate < 130 or > 50 beats/minute
* Peripheral pulse oxygen saturation > 90%
* Arterial oxygen partial pressure (PaO2) ≥ 70 mmHg
* Arterial pH ≥ 7.25.

Administration of contrast agent Sonovue requires an infusion pump (Vueject, Bracco, Milan, Italy), which provides constant agitation to maintain the homogeneity distribution of Sonovue. Injection of Sonovue allows an enhancement of LV endocardial border and regional function to evaluate:

* LV end-diastolic and end-systolic volumes (ml) and ejection fraction (%) using the Simpson method.
* The WMSI of the left ventricle (LV) after Sonovue injection.

After optimization of transthoracic cardiac views, the mechanical index will settle between 0.1-0.2 and keeps unchanged during the procedure. Sonovue vial of 5 ml will dilute in in 10 ml saline solution and administrate at 0.7-1.5 ml/min. Using acquire flash-replenishment sequences during15 cardiac cycles of the apical 4-2-3 chamber views with the flash delivered after the second cardiac cycle. This technique destroys the microbubbles presents in the myocardium and allows replenishment with new microbubbles concentrations.

The volume of blood within the entire coronary circulation at rest in diastole is predominantly resided within the capillaries. The myocardial signal intensity emanating from the contrast agent reflects the concentration of microbubbles within the myocardium. It takes 5 seconds for complete replenishment of the myocardium. Any decrease in myocardial blood flow prolongs replenishment time in proportion to its reduction.

Immediately after microbubble infusion is started, all real-time MCE procedures are recorded for one minute and stored as DICOM (Digital Image Communications in Medicine) images. Offline analysis uses a specific quantification software named QLAB10 (Philips Medical Systems, the Netherlands) to convert myocardial perfusion images into time-intensity curves (TIC) corresponding to different regions of interest (ROI) of the 16 myocardial segments.

Four variables are analyzed from these TIC curves to evaluate qualitatively the myocardial microcirculation:

* peak intensity (PI) in decibel (dB).
* time to peak intensity in seconds (TTP).
* mean transit time in seconds (MTT).
* Area under the curve in dB/seconds (AUC).

The cardiac biomarkers including High sensivity cardiac troponin I for myocardial injury and N-terminal pro-brain natriuretic peptide (NT-proBNP) for heart failure are measured once daily in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis: a life-threatening organ dysfunction (defined as an acute change in total Sequential Organ Failure Assessment (SOFA) score > 2 points consequent to infection) caused by a dysregulated host response to infection.
* Sepsis shock : a subset of sepsis with persisting hypotension requiring vasopressors to maintain the mean arterial pressure > 65 mmHg and having a serum lactate level > 2 mmol/L after fluid resuscitation.

Exclusion Criteria:

* Non-survivors in the first 24 hours from sepsis
* Sepsis post-acute cardiac arrest
* Pregnancy
* Younger than 18 years old
* Acute Respiratory Distress Syndrome (ARDS) with the ratio of arterial oxygen partial pressure (mmHg) to fractional inspired oxygen (PaO2/ FiO2) < 200)
* Advanced malignancy
* Untreated and unstable acute coronary syndrome
* History of myocardial infarction with severe left ventricular dysfunction. (Ejection fraction < 20 %).
* Inoperable valvular and coronary disease
* Significant right-left cardiac shunt
* Untreated congenital heart disease
* Severe systolic pulmonary hypertension > 80 mmHg
* Insufficient echogenicity
* Prior anaphylaxis reaction to the Sonovue microbubbles

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of the time to Peak intensity (TTP) from baseline (seconds). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Qualitative evaluation of myocardial microcirculation using the variables of the time-intensity curve after Sonovue administration: The investigators hypothesize that patients who develop cardiac dysfunction will have a prolonged time to Peak intensity over time.
Mean change of the Mean transit time (MTT) from baseline (seconds) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Qualitative evaluation of myocardial microcirculation using the variables of the time-intensity curve after Sonovue administration: The investigators hypothesize that patients who develop cardiac dysfunction will have a prolonged Mean transit time over time.
Mean change of the Peak intensity (PI) from baseline (seconds). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Qualitative evaluation of myocardial microcirculation using the variables of the time-intensity curve after Sonovue administration: The investigators hypothesize that patients who develop cardiac dysfunction will have a reduced Peak intensity over time
Mean change of the Area under the curve (AUC) from baseline (dB/ seconds). | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Qualitative evaluation of myocardial microcirculation using the variables of the time-intensity curve after Sonovue administration: The investigators hypothesize that patients who develop cardiac dysfunction will have a reduced Area under the curve (AUC) over time
Mean change of the Wall motion score index (WMSI) from baseline (normal score: 32) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Quantitative evaluation of the regional contractility of 16 myocardial segments of LV using the Wall motion score index. The investigators expect a lower score than 32 in patients who develop cardiac dysfunction over time
Mean change of the ejection fraction from baseline (%) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Quantitative evaluation of the global LV ejection fraction using the Simpson method. The investigators expect a lower ejection fraction than 50% in patients who develop cardiac dysfunction over time.
Mean change of the Tricuspid annular plane systolic excursion (TAPSE) of the right ventricle from baseline (mm) | Comparison to baseline (24 hours after ICU admission) to the two other time points: at 48 to 72 hours, at 5 to 10 days after withdrawal of vasopressor and inotropic agents.
  Quantitative evaluation of the longitudinal contractility of the right ventricle by measuring the Tricuspid annular plane systolic excursion (TAPSE) with pulsed tissue doppler. The investigators expect lower values than 15 mm in patients who develop cardiac dysfunction over time.

SECONDARY OUTCOMES:
Mean change of biomarker of cardiac injury: serum High sensitivity cardiac troponin I (micrograms/ L) from baseline. | Comparison to baseline (24 hours after ICU admission) and then once daily during the study period
  Evaluation of the severity of myocardial injury associated with cardiac dysfunction by measuring High sensitivity cardiac troponin I. The investigators expect patients who develop cardiac dysfunction will have higher serum levels of this biomarker than those who do not over time.
Mean change of biomarker of heart failure: serum N-terminal pro-brain natriuretic peptide (NT-proBNP) (nanograms/ L) from baseline. | Comparison to baseline (24 hours after ICU admission) and then once daily during the study period
  Evaluation of the degree of heart failure associated with cardiac dysfunction by measuring N-terminal pro-brain natriuretic peptide (NT-proBNP). The investigators expect patients who develop cardiac dysfunction will have higher serum levels of this biomarker than those who do not over time.

CONTACTS AND LOCATIONS:
Overall Officials: Duc Nam Nguyen, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senior R, Becher H, Monaghan M, Agati L, Zamorano J, Vanoverschelde JL, Nihoyannopoulos P, Edvardsen T, Lancellotti P; EACVI Scientific Documents Committee for 2014-16 and 2016-18; EACVI Scientific Documents Committee for 2014-16 and 2016-18. Clinical practice of contrast echocardiography: recommendation by the European Association of Cardiovascular Imaging (EACVI) 2017. Eur Heart J Cardiovasc Imaging. 2017 Nov 1;18(11):1205-1205af. doi: 10.1093/ehjci/jex182. PMID 28950366
- [Background] Orde S, McLean A. Bedside myocardial perfusion assessment with contrast echocardiography. Crit Care. 2016 Mar 15;20:58. doi: 10.1186/s13054-016-1215-7. PMID 26976127
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise J, Solomon S, Spencer KT, St John Sutton M, Stewart W; American Society of Echocardiography's Nomenclature and Standards Committee; Task Force on Chamber Quantification; American College of Cardiology Echocardiography Committee; American Heart Association; European Association of Echocardiography, European Society of Cardiology. Recommendations for chamber quantification. Eur J Echocardiogr. 2006 Mar;7(2):79-108. doi: 10.1016/j.euje.2005.12.014. Epub 2006 Feb 2. PMID 16458610
- [Background] Beesley SJ, Weber G, Sarge T, Nikravan S, Grissom CK, Lanspa MJ, Shahul S, Brown SM. Septic Cardiomyopathy. Crit Care Med. 2018 Apr;46(4):625-634. doi: 10.1097/CCM.0000000000002851. PMID 29227368